CLINICAL TRIAL: NCT06428955
Title: Prospective Multicenter Evaluation of the Visual Performance of a Non-constant Aberration Correcting Aspheric Monofocal Intraocular Lens (Precise Study)
Brief Title: Evaluation of a Monofocal Intraocular Lens
Acronym: PRECISE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GPAS-SAS-023-01
Record Dates: First submitted 2024-05-15; First posted 2024-05-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Bilateral implantation of investigational device (Experimental): Monofocal IOL
  Interventions: Device: CT LUCIA 621P

INTERVENTIONS:
Device: CT LUCIA 621P — The device under investigation, CT LUCIA 621P IOL (Carl Zeiss Meditec, Jena, Germany) is a posterior chamber intraocular lens which is indicated for aphakia after surgical extraction of the cataractous natural lens. It is a monofocal aspheric IOL made of hydrophobic material and coated with heparin. The modified C-loop haptic is step-vaulted.

SUMMARY:
The aim of this study is to investigate the 3-month visual performance of the CT LUCIA 621P IOL, a hydrophobic aspheric monofocal IOL with a non-constant aspheric optic profile in adult patients 50 years of age or older who are undergoing cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 50 years of age or older, male or female, of any race or ethnicity.
2. Presenting for uncomplicated bilateral cataract surgery for age-related cataract.
3. Planned bilateral cataract extraction with posterior chamber IOL implantation, via phacoemulsification with or without femtosecond laser assisted cataract surgery (FLACS).
4. Bilateral implantation of a CT LUCIA 621P IOL with a dioptric power between +10.00 D and +30.00 D and a target postoperative refraction of emmetropia (0.00 ±0.50 D).
5. Clear intraocular media other than cataract (i.e. no hyphema, vitreous hemorrhage)
6. No visual acuity limiting pathologies other than cataract. Best corrected postoperative visual acuity potential of 20/25 or better in both eyes as estimated by potential acuity meter or surgeon estimation.
7. Provide written informed consent and a signed HIPPA form.
8. Availability, willingness, ability, and sufficient cognitive awareness to comply with study examination procedures and the schedule for study visits and evaluations.

Exclusion Criteria:

1. Corneal Astigmatism of >1.0 D.
2. Planned monocular cataract extraction.
3. Visual field loss which has an impact on visual acuity.
4. Subjects with intraoperative surgical complications in whom a CT LUCIA 621P IOL cannot be implanted.
5. History of acute or chronic disease, pathology, illness, or ocular trauma that would, in the surgeon's opinion, confound results (e.g., corneal pathology, keratoconus, strabismus, uncontrolled glaucoma)
6. History of Glaucoma, macular degeneration, cystoid macular edema, proliferative diabetic retinopathy, amblyopia, etc.
7. Previous intraocular or corneal surgery, including all forms of refractive surgery that might confound the outcome of the investigation or increase the risk to the subject
8. Previous anterior or posterior chamber surgery other than peripheral retinal barrier laser, SLT/ALT (e.g., vitrectomy, laser iridotomy)
9. Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils or pupils that do not dilate under mesopic/scotopic conditions).
10. Capsular or zonular abnormalities or other conditions that increase the risk of zonular rupture during cataract extraction procedure and/or may affect the postoperative centration or tilt of the lens
11. Use of a systemic or ocular medication that might affect vision and confound the outcome or increase the risk to the subject in the opinion of the investigator such as tamsulosin hydrochloride (Flomax) or other medications with similar side effects (floppy iris syndrome)
12. Cycloplegic pupil diameter <6.0 mm or the presence of ocular implants that limit pupil diameter (malyugin rings; iris prosthesis).
13. Usage of contact lenses during study participation
14. Pregnant, lactating during the course of the investigation, or has another condition with associated fluctuation of hormones that could lead to refractive changes
15. Presence or history or any other condition or finding that, in the investigator's opinion, makes the subject unsuitable as a candidate for study participation, may increase the operative risk or may confound the outcome of the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Monocular best corrected distance visual acuity (CDVA) | Three (3) Months
  The primary efficacy endpoint is the proportion of patients with monocular CDVA of 20/40 or better at three months

SECONDARY OUTCOMES:
Binocular Corrected Distance Visual Acuity | Three (3) Months
Monocular Uncorrected Distance Visual Acuity | Three (3) Months
Monocular Distance Corrected Intermediate Visual Acuity | Three (3) Months
Monocular Uncorrected Intermediate Visual Acuity | Three (3) Months
Manifest Refraction Spherical Equivalent | Three (3) Months
Refractive Predictability | Three (3) Months
  Manifest refraction will be evaluated at 1 and 3 months to determine refractive predictability. The predicted refraction is the goal or target refraction from the IOLMaster IOL calculation and the observed refraction is the 3 Month postoperative Manifest Refraction Spherical Equivalent measurement.
Refractive Stability | Three (3) Months
  Manifest refraction will be obtained at 1 and 3 months to evaluate whether refractive stability is achieved by 3 months. Refractive stability will be evaluated at the 1 to 3 months interval as a parameter of interest to determine the proportion of eyes that achieve stability of manifest refraction.
Contrast Sensitivity - mesopic and photopic with and without glare | Three (3) Months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Price Vision Group, Indianapolis, Indiana
  - Huffman & Huffman PSC, Lexington, Kentucky
  - The Pennsylvania State University and Penn State Health, Hershey, Pennsylvania
- Asociación Para Evitar La Ceguera en México, I.A.P., Mexico City, Alcaldia Coyoacan, Mexico

IPD SHARING:
Plan to Share IPD: No